CLINICAL TRIAL: NCT04651972
Title: Diagnostic of Autism by Measurement of vanilloïd Compounds in Urin
Brief Title: Measurement of vanilloïd Compounds in Urin of Autistic vs Control Patients, as Potential Biomarkers
Acronym: DIADAUVEDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Marc MERTEN, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2020PI116
Record Dates: First submitted 2020-10-05; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — urines
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a former study, four vanilloid compounds were observed increased in the urin of autistic patients. The present study is aimed at performing a ambispective study to confirm or not these preliminary results. 70 urins from autistic children (already collected) will be compared to 70 urins of non autistic children (collected without intervention, remaining sample from the standard care), in terms of measurements of four vanilloid compounds using a GCMS apparatus.

ELIGIBILITY:
Inclusion criteria :

For cases :

* Male children aged 2 years to less than 15 years inclusive years at time of sample collection
* Children with a diagnosis of autism (ICD-10 F84.0) after assessment by a child psychiatrist.

For healthy chlidren:

* Children aged 2 years to less than 15 years old performing an ECBU at the CHRU of Nancy as part of their care.
* Patient whose ECBU is negative with respect to cytobacteriology (absence of urinary infection).
* Child can be matched to a CAS

Exclusion criteria

For cases:

* Children in whom one of the following pathologies is found during the anamnesis or in the clinical record : (i) renal insufficiency; (ii) urinary tract infection at the time of sampling and/or metabolic disease
* Children on antibiotic treatment at the time of collection

For healthy chlidren :

* children whose urine culture come from one of the following departments: Pediatric Nephrology (potential risk of renal failure) or Pediatric Neurology (potential risk of neurological disorder).
* with a diagnosis of autism
* with a metabolic disease
* children undergoing antibiotic treatment at the time of collectio

Ages: 2 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — only males will be studied
Study Population: Autistic children according to CM-10 (F84.0)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
measurements of vanilloid compound in urins | through study completion, an average of 18 months
  The primary end point is to determine if isolated or combinations of vanilloid compound measured in urin, may discriminate autistic vs non autistic childen

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Olivier, MD, PhD,, Study Director — CHRU Nancy